CLINICAL TRIAL: NCT00666757
Title: TRY FIRST: A 12-Week, Randomized, Open-Label Trial of Duloxetine Versus Generic SSRIs in the Treatment of a Severe Depressive Episode
Brief Title: A Study Comparing Duloxetine to Other Antidepressants in the Treatment of Severe Depression
Acronym: TRY FIRST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11715; F1J-US-HMFT (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Results first posted 2010-06-15 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2010-05

CONDITIONS: Depression
Keywords: Severe Depressive Episode
MeSH Terms: conditions — Depression | interventions — Duloxetine Hydrochloride; Fluoxetine; Citalopram; Paroxetine; Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- duloxetine (Experimental): study drug
  Interventions: Drug: duloxetine
- citalopram (Active Comparator)
  Interventions: Drug: citalopram
- fluoxetine (Active Comparator)
  Interventions: Drug: fluoxetine
- paroxetine (Active Comparator)
  Interventions: Drug: paroxetine
- sertraline (Active Comparator)
  Interventions: Drug: sertraline

INTERVENTIONS:
Drug: duloxetine — 30-120 milligrams (mgs) orally daily for 12 weeks
  Other Names: LY248686; Cymbalta
  Arms: duloxetine
Drug: fluoxetine — 20-80 mgs orally daily for 12 weeks
  Arms: fluoxetine
Drug: citalopram — 20-40 mgs orally daily for 12 weeks
  Arms: citalopram
Drug: paroxetine — 20-50 mgs orally daily for 12 weeks
  Arms: paroxetine
Drug: sertraline — 50-200 mgs orally daily for 12 weeks
  Arms: sertraline

SUMMARY:
The purpose of this study is to compare duloxetine with other antidepressants in the treatment of severe depression.

ELIGIBILITY:
Inclusion criteria:

* At least 18 years of age
* Have major depression and are currently in a severe depressive episode
* Have a degree of understanding such that patient can communicate with the investigator and study staff
* All females must test negative for pregnancy
* Females of childbearing potential must use reliable method of birth control during the study and for 1 month after taking the last dose of study drug

Exclusion criteria:

* Have not responded to duloxetine for depression in the past
* Have a history of bipolar disorder, a psychotic disorder (such as schizophrenia), a cognitive disorder (such as moderate or severe dementia), or obsessive-compulsive disorder (OCD)
* Are at significant risk for suicide
* Have not responded to 2 or more adequate trials of antidepressant medications during the current depressive episode
* Have a serious, unstable medical condition
* Have a current or recent history of substance abuse or dependence
* Have had electroconvulsive therapy (ECT), transcranial magnetic stimulation (rTMS), or vagus nerve stimulation (VNS) in the past year
* Have started psychotherapy within 6 weeks prior to study entry
* Have a serious medical illness or clinically significant laboratory abnormality that is not stabilized or is anticipated, in the judgment of the investigator, to require hospitalization or use of an excluded medication during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2008-05; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5PM Eastern Time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (61):
- United States (61):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carson, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Irvine, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherman Oaks, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torrance, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pueblo, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clearwater, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coral Springs, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Deerfield Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hialeah, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melbourne, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winter Park, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Joliet, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oak Brook, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Park Ridge, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenwood, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Terre Haute, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prairie Village, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gaithersburg, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glen Burnie, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rockville, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fall River, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clementon, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Princeton, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresh Meadows, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mount Kisco, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beachwood, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dayton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kettering, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eugene, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Havertown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Media, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newtown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lincoln, Rhode Island
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sioux Falls, South Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Friendswood, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Jackson, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita Falls, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Woodstock, Vermont
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlottesville, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herndon, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellevue, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brown Deer, Wisconsin

REFERENCES:
- [Derived] Dodd S, Berk M, Kelin K, Zhang Q, Eriksson E, Deberdt W, Craig Nelson J. Application of the Gradient Boosted method in randomised clinical trials: Participant variables that contribute to depression treatment efficacy of duloxetine, SSRIs or placebo. J Affect Disord. 2014 Oct;168:284-93. doi: 10.1016/j.jad.2014.05.014. Epub 2014 Jun 4. PMID 25080392
- [Derived] Martinez JM, Katon W, Greist JH, Kroenke K, Thase ME, Meyers AL, Edwards SE, Marangell LB, Shoemaker S, Swindle R. A pragmatic 12-week, randomized trial of duloxetine versus generic selective serotonin-reuptake inhibitors in the treatment of adult outpatients in a moderate-to-severe depressive episode. Int Clin Psychopharmacol. 2012 Jan;27(1):17-26. doi: 10.1097/YIC.0b013e32834ce11b. PMID 22027844
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The United States study started in May 2008 and completed in March 2009. A total of 72 sites participated (65 Psychiatric, 5 Family Practice, and 2 Internal Medicine specialties).
Groups:
- Selective Serotonin Reuptake Inhibitor (SSRI): all comparator SSRIs pooled together: citalopram 20-40 mgs orally daily for 12 weeks; fluoxetine 20-80 mg orally daily for 12 weeks; paroxetine 20-50 mgs orally daily for 12 weeks; and sertraline 50-200 mgs orally daily for 12 weeks
Period: Overall Study
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Started | 372 | 378
Completed | 272 | 281
Not Completed | 100 | 97
Not completed — Lost to Follow-up | 39 | 35
Not completed — Protocol Violation | 23 | 24
Not completed — Adverse Event | 22 | 12
Not completed — Withdrawal by Subject | 13 | 17
Not completed — Lack of Efficacy | 3 | 6
Not completed — Physician Decision | 0 | 2
Not completed — Sponsor decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI) | Total
Number analyzed (Participants) | 372 | 378 | 750
Age Continuous [Mean (Standard Deviation); unit: years] | 44.3 (13.01) | 43.8 (13.05) | 44.1 (13.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 237 | 259 | 496
  Male | 135 | 119 | 254
Race/Ethnicity, Customized [Number; unit: participants]
  African Descent | 76 | 68 | 144
  Caucasian | 231 | 241 | 472
  East/Southeast Asian | 2 | 7 | 9
  Hispanic | 59 | 52 | 111
  Western Asian | 1 | 2 | 3
  Other | 3 | 7 | 10
  Missing | 0 | 1 | 1
Region of Enrollment [Number; unit: participants] — United States study
  participants
    United States | 372 | 378 | 750
History, Met Diagnosis of Major Mood Disorder (MDD) [Number; unit: participants] | 372 | 378 | 750
17-Item Hamilton Depression Rating Scale (HAMD-17) Anxiety/Somatization Subscale Score [Mean (Standard Deviation); unit: units on a scale] — HAMD-17 Anxiety/Somatization subscale consists of items 10, 11, 12, 13, 15, and 17 evaluates agitation, and severity of psychic and somatic manifestations of anxiety. Total subscale scores range from 0 (normal) to 18 (severe).
  units on a scale | 7.45 (2.22) | 7.42 (2.25) | 7.43 (2.23)
17-Item Hamilton Depression Rating Scale (HAMD-17) Bech Subscale Score [Mean (Standard Deviation); unit: units on a scale] — HAMD-17 Bech subscale consists of items 1, 2, 7, 8, 10, and 13 used to evaluate core symptoms of Major Depressive Disorder (MDD). Total subscale scores range from 0 (normal) to 22 (severe).
  units on a scale | 12.97 (2.13) | 13.13 (1.95) | 13.05 (2.04)
17-Item Hamilton Depression Rating Scale (HAMD-17) Maier Subscale Score [Mean (Standard Deviation); unit: units on a scale] — HAMD-17 Maier Subscale consists of Items 1, 2, 7, 8, 9, 10 and represents the "core" symptoms of depression. Total subscale scores range from 0 (normal) to 24 (severe).
  units on a scale | 12.47 (2.33) | 12.48 (2.22) | 12.47 (2.27)
17-Item Hamilton Depression Rating Scale (HAMD-17) Retardation Subscale [Mean (Standard Deviation); unit: units on a scale] — The HAMD-17 Retardation subscale consists of Items 1, 7, 8, 14 and evaluates dysfunction in mood, work, and sexual activity, as well as overall motor retardation. Total subscale scores range from 0 (normal) to 14 (severe).
  units on a scale | 8.36 (1.55) | 8.53 (1.54) | 8.45 (1.55)
17-Item Hamilton Depression Rating Scale (HAMD-17) Sleep Subscale Score [Mean (Standard Deviation); unit: units on a scale] — The HAMD-17 Sleep Subscale consists of Items 4, 5, 6 and evaluates initial, middle, and late insomnia. Total subscale scores range from 0 (no difficulty) to 6 (difficulty).
  units on a scale | 4.73 (1.35) | 4.77 (1.33) | 4.75 (1.34)
17-Item Hamilton Depression Rating Scale (HAMD-17) Total Score [Mean (Standard Deviation); unit: units on a scale] — The HAMD-17 Total Score is a rater-administered assessment of depression severity and improvement, with total score ranges from 0 (not at all depressed) to 52 (most severely depressed).
  units on a scale | 25.03 (4.44) | 25.03 (4.24) | 25.03 (4.34)
Brief Pain Inventory (BPI) Average 24-Hour Pain Score [Mean (Standard Deviation); unit: units on a scale] — The BPI is a self-reported scale measuring pain severity and pain-specific interference on function on a scale ranging from 0 (no pain) to 10 (pain as bad as you can imagine).
  units on a scale | 2.64 (2.74) | 2.98 (2.79) | 2.81 (2.77)
History, Age at First Episode [Mean (Standard Deviation); unit: years] — Age when first MDD episode occurred
  years | 31.53 (14.39) | 30.42 (14.30) | 30.97 (14.34)
History, Number of Previous MDD Episodes [Mean (Standard Deviation); unit: episodes] — Number of previous MDD episodes
  episodes | 6.74 (15.32) | 5.09 (11.08) | 5.91 (13.37)
History, Time Since Most Recent MDD Episode [Mean (Standard Deviation); unit: months] — Number of months since most recent MDD episode
  months | 11.76 (19.06) | 11.92 (30.69) | 11.84 (25.57)
Quick Inventory of Depressive Symptomatology (QIDS-SR) Total Score [Mean (Standard Deviation); unit: units on a scale] — The QIDS-SR Total Score is a 16-item, participant-rated short form of the Inventory of Depressive Symptomatology that assesses 9 domains: sad mood, concentration, self-outlook, suicidal ideation, involvement, energy/fatigability, sleep disturbance, appetite/weight increase/decrease and psychomotor agitation/retardation. Scores range from 0 (none) to 27 (very severe) depression.
  units on a scale | 21.64 (1.71) | 21.70 (1.70) | 21.67 (1.701)
Sheehan Disability Scale (SDS) Global Functional Impairment Score [Mean (Standard Deviation); unit: units on a scale] — The SDS Global Functional Impairment Score is a total score that is calculated by summing the SDS Item 1, 2, and 3; the score ranges from 0 (unimpaired) to 30 (highly impaired).
  units on a scale | 22.70 (5.52) | 22.72 (6.05) | 22.71 (5.79)
Sheehan Disability Scale (SDS) Item 1: Symptoms Disrupted Work/School [Mean (Standard Deviation); unit: units on a scale] — The SDS is completed by the participant and Item 1 is used to assess the effect of the participant's symptoms on their work/school schedule. Scores range from 0 to 10 with higher values indicating greater disruption in the participant's work/school life.
  units on a scale | 7.00 (2.40) | 7.09 (2.45) | 7.05 (2.42)
Sheehan Disability Scale (SDS) Item 2: Symptoms Disrupted Social Life/Leisure Activities [Mean (Standard Deviation); unit: units on a scale] — The SDS is completed by the participant and is used to assess the effect of the participant's symptoms on their work/social/family life. Total scores range from 0 to 30 with higher values indicating greater disruption in the participant's work/social/family life.
  units on a scale | 7.81 (1.97) | 7.82 (2.13) | 7.82 (2.05)
Sheehan Disability Scale (SDS) Item 3: Symptoms Disrupted Family Life/Home Responsibilities [Mean (Standard Deviation); unit: units on a scale] — The SDS is completed by the participant and Item 3 is used to assess the effect of the participant's symptoms on their family life/home responsibilities. Scores range from 0 to 10 with higher values indicating greater disruption in the participant's family life/home responsibilities.
  units on a scale | 7.67 (2.02) | 7.68 (2.28) | 7.67 (2.15)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 86.62 (22.37) | 86.23 (23.97) | 86.42 (23.18)
World Health Organization Health and Work Performance Questionnaire (HPQ), Absolute Absenteeism [Mean (Standard Deviation); unit: hours lost per week] — The HPQ was used to assess the total hours of missed work (absenteeism) per week. The calculation for absolute absenteeism is actual hours worked minus expected hours equals number of missed work days.
  hours lost per week | 28.64 (59.28) | 33.29 (72.90) | 31.00 (66.48)
World Health Organization Health and Work Performance Questionnaire (HPQ), Absolute Presenteeism [Mean (Standard Deviation); unit: units on a scale] — The HPQ was used to assess the participant's performance at work. Participants rated their overall performance on the days worked in the last week on a scale of 0 (worst performance) to 10 (top performance). Values were then multiplied by 10 to create a percentage scale between 0 and 100 percent. Absolute presenteeism equals the difference between the "score for self" and "score for average worker in same job".
  units on a scale | 48.85 (22.47) | 50.63 (23.86) | 49.74 (23.16)

OUTCOME MEASURES:

1. Primary Outcome: Probability of Remission [16-item Quick Inventory of Depressive Symptomatology (QIDS-SR) Score Less Than or Equal to 5 at 12-Week Endpoint]
Description: Visitwise probability of participants per treatment meeting remission criteria (QIDS-SR total score [TS]</=5 at week 12 endpoint) were estimated using a pseudolikelihood-based mixed-models repeated measures analysis for a categorical outcome, model included fixed, categorical effects of treatment group (duloxetine vs. SSRIs), visit, treatment group-by-visit & continuous, fixed covariate of baseline QIDS-SR TS, and random effect of participant. Primary analysis contrasted remission probability at week 12 endpoint between treatment groups.
Time Frame: 12 weeks
Population: Intent to Treat. Data based on number of subjects enrolled at Week 0: Duloxetine N=366, SSRI N=371; and Week 12: Duloxetine N=273, SSRI N=284
Measure: Least Squares Mean (Standard Error); unit: Probability of remission
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 273 | 284
Probability of remission | 0.36 (0.03) | 0.32 (0.03)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); Categorical, pseudo-likelihood-based repeated measures approach (MMRM-CAT). The analysis will contrast the remission rates at 12 week endpoint between treatment groups; Test type: Superiority or Other; p = 0.26, Mixed Models Analysis

2. Secondary Outcome: Change From Baseline in QIDS-SR Total Score at 12-Week Endpoint (Mood Measure)
Description: The QIDS-SR is a 16-item, participant-rated short form of the Inventory of Depressive Symptomatology that assesses 9 domains: sad mood, concentration, self-outlook, suicidal ideation, involvement, energy/fatigability, sleep disturbance, appetite/weight increase/decrease and psychomotor agitation/retardation. Scores range from 0 (none) to 27 (very severe). The QIDS-SR total score was used to derive the mean change from baseline to endpoint depression.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 273 | 284
units on a scale | -13.4 (0.36) | -12.6 (0.35)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); Repeated Measures Analysis.Treatment comparisons will include the contrast between treatment groups at 12-week endpoint; Test type: Superiority or Other; p = 0.07, Mixed Models Analysis

3. Secondary Outcome: Probability of Remission [17-item Hamilton Depression Rating Scale (HAMD-17) (Mood Measure) Less Than or Equal to 7 at 12-Week Endpoint]
Description: Visitwise percentages of participants meeting remission criteria HAMD-17 total score [TS] </=7 at week 12 endpoint) were estimated using a categorical, pseudolike-lihood-based repeated measures approach, & included fixed, categorical effects of treatment group (duloxetine vs. SSRIs), visit, treatment group-by-visit interaction, & continuous, fixed covariate of baseline HAMD-17 TS. Primary analysis will be contrast of remission rates at week 12 endpoint between treatment groups, & represents estimated remission rates for each treatment group had all participants completed 12 weeks of therapy.
Time Frame: 12 weeks
Population: Intent to treat. Data based on number of subjects enrolled at Week 0: Duloxetine N=365, SSRI N=371 and Week 12: Duloxetine N=272, SSRI N=283
Measure: Least Squares Mean (Standard Error); unit: Probability of remission
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 272 | 283
Probability of remission | 0.53 (0.03) | 0.44 (0.03)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); Categorical, pseudo-likelihood-based repeated measures approach (MMRM-CAT). Repeated Measures Analysis. The analysis will contrast the remission remission rates at 12-week endpoint; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis

4. Secondary Outcome: Probability of Response [QIDS-SR Total Score (Mood Measure) Greater Than Or Equal To 50 Percent Reduction From Baseline To 12 Week Endpoint]
Description: Visitwise percentages of participants meeting response criteria (50% reduction from baseline QIDS-SR total score at 12-week endpoint) were estimated using a categorical, pseudolikelihood-based repeated measures approach, & included fixed, categorical effects of treatment group, visit, treatment group-by-visit interaction, & continuous, fixed covariate of baseline QIDS-SR. The primary analysis will be the contrast of response rates at week 12 endpoint between treatment groups, and represents estimated response rates for each treatment group had all participants completed 12 weeks of therapy.
Time Frame: Baseline, 12-Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Probability of response
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 273 | 284
Probability of response | 0.71 (0.03) | 0.64 (0.03)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); Categorical, pseudo-likelihood-based repeated measures approach (MMRM-CAT). The analysis will contrast the response rates at 12-week endpoint; Test type: Superiority or Other; p = 0.09, Mixed Models Analysis

5. Secondary Outcome: Probability of Response [HAMD-17 Total Score (Mood Measure) Greater Than Or Equal To 50 Percent Reduction From Baseline To 12 Week Endpoint]
Description: Visitwise percentages of participants meeting response criteria 50% reduction from baseline in HAMD-17 total score at 12-Week endpoint) were estimated using a categorical, pseudolike-lihood-based repeated measures approach, & included fixed, categorical effects of treatment group, visit, treatment group-by-visit interaction, & continuous, fixed covariate of baseline HAMD-17 TS. Primary analysis will be the contrast of response rates at week 12 endpoint between treatment groups, & represents estimated response rates for each treatment group had all participants completed 12 weeks of therapy.
Time Frame: Baseline, 12-Weeks
Population: Intent to treat. Data based on number of subjects enrolled at Week 0: Duloxetine N=365, SSRI N=371; and Week 12: Duloxetine N=272, SSRI N=283
Measure: Least Squares Mean (Standard Error); unit: Probability of response
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 272 | 283
Probability of response | 0.73 (0.03) | 0.61 (0.03)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis

6. Secondary Outcome: Change From Baseline in HAMD-17 Total Score at 12-Week Endpoint (Mood Measure)
Description: The HAMD-17 is a rater-administered assessment of depression severity and improvement, with total score ranges from 0 (not at all depressed) to 52 (most severely depressed).
Time Frame: Baseline, 12 Weeks
Population: Intent to Treat. Data based on number of subjects enrolled at Week 0: Duloxetine N=365, SSRI N=371; and; and Week 12: Duloxetine N=272, SSRI N=283
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 272 | 283
units on a scale | -17.03 (0.43) | -15.3 (0.42)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); Repeated Measures Analysis. Treatment comparisons will include the contrast between treatment groups at 12-Week endpoint; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis

7. Secondary Outcome: Change From Baseline in HAMD-17 Anxiety/Somatization Subscale Score at 12-Week Endpoint (Mood Measure)
Description: HAMD-17 subscale consists of items 10, 11, 12, 13, 15, and 17 evaluates agitation, and severity of psychic and somatic manifestations of anxiety. Total subscale scores range from 0 (normal) to 18 (severe). Mean change from baseline to endpoint.
Time Frame: Baseline, 12 Weeks
Population: Intent to Treat. Data based on number of subjects enrolled at Week 0: Duloxetine N=367, SSRI N=371; and Week 12: Duloxetine N=274, SSRI N=284
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 274 | 284
units on a scale | -4.89 (0.16) | -4.24 (0.15)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis

8. Secondary Outcome: Change From Baseline in HAMD-17 Maier Subscale Score at 12-Week Endpoint (Mood Measure)
Description: HAMD-17 Maier Subscale consists of Items 1, 2, 7, 8, 9, 10 and represents the "core" symptoms of depression. Total subscale scores range from 0 (normal) to 24 (severe).
Time Frame: Baseline, 12 weeks
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 274 | 284
units on a scale | -9.01 (0.23) | -8.16 (0.22)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis

9. Secondary Outcome: Change From Baseline in HAMD-17 Bech Subscale Score at 12-Week Endpoint (Mood Measure)
Description: HAMD-17 Bech subscale consists of items 1, 2, 7, 8, 10, and 13 used to evaluate core symptoms of Major Depressive Disorder (MDD). Total subscale scores range from 0 (normal) to 22 (severe).
Time Frame: Baseline, 12 Weeks
Population: Intent to Treat. Data based on number of subjects enrolled at Week 0: Duloxetine N=367, SSRI N=371; and Week 12: Duloxetine N=274; SSRI N=284
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 274 | 284
units on a scale | -9.21 (0.24) | -8.40 (0.24)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); Repeated Measures Analysis.Treatment comparisons will include the contrast between treatment groups at 12-Week endpoint; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis

10. Secondary Outcome: Change From Baseline in HAMD-17 Retardation Subscale Score at 12-Week Endpoint (Mood Measure)
Description: The HAMD-17 Retardation subscale consists of Items 1, 7, 8, 14 and evaluates dysfunction in mood, work, and sexual activity, as well as overall motor retardation. Total subscale scores range from 0 (normal) to 14 (severe).
Time Frame: Baseline, 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 273 | 284
units on a scale | -5.99 (0.16) | -5.49 (0.16)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis

11. Secondary Outcome: Change From Baseline in HAMD-17 Sleep Subscale Score at 12-Week Endpoint (Mood Measure)
Description: The HAMD-17 Sleep Subscale consists of Items 4, 5, 6 and evaluates initial, middle, and late insomnia. Total subscale scores range from 0 (no difficulty) to 6 (difficulty).
Time Frame: Baseline, 12 Weeks
Population: Intent to Treat. Data based on number of subjects enrolled at Week 0: Duloxetine N=367, SSRI N=371; and Week 12: Duloxetine N=274, SSRI N=285
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 274 | 285
units on a scale | -2.77 (0.12) | -2.58 (0.12)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.20, Mixed Models Analysis

12. Secondary Outcome: Change From Baseline in Brief Pain Inventory (BPI) Average 24-hour Pain Score, in Particpants With a Baseline BPI Average 24-hour Pain Score of 3 or Greater, at 12-Week Endpoint (Pain Measure)
Description: The BPI is a self-reported scale measuring pain severity and pain-specific interference on function on a scale ranging from 0 (no pain) to 10 (pain as bad as you can imagine). The BPI average 24-hour pain measure was used to derive the overall mean change from baseline to endpoint, in those participants who had a BPI average 24-hour pain score of 3 or greater at baseline.
Time Frame: Baseline, 12 Weeks
Population: Intent to Treat. Data based on number of subjects enrolled at Week 0: Duloxetine N=211, SSRI N=233; and Week 12: Duloxetine N=156, N=166
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 156 | 166
units on a scale | -2.95 (0.21) | -2.39 (0.20)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); Only those patients who had at least moderate pain at baseline (defined as baseline BPI Average 24-Hour Pain Score greater than or equal to 3). Repeated Measures Analysis. Treatment comparisons will include the contrast between treatment groups at 12-Week endpoint; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis

13. Secondary Outcome: Change From Baseline in BPI Average 24 Hour Pain Score at 12-Week Endpoint (Pain Measure)
Description: The BPI is a self-reported scale measuring pain severity and pain-specific interference on function, with scores ranging from 0 (does not interfere) to 10 (completely interferes). The BPI average 24-hour pain measure was used to derive the overall mean change from baseline to endpoint.
Time Frame: Baseline, 12 weeks
Population: Intent to Treat. Data based on number of subjects enrolled at Week 0: Duloxetine N=346, SSRI N=348; and Week 12: Duloxetine N=249, SSRI N=257
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 249 | 257
units on a scale | -1.83 (0.15) | -1.43 (0.15)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis

14. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Global Functional Impairment Score at 12-Week Endpoint (Functional Outcome Measure)
Description: The SDS is a participant-rated anchored visual analog scale to assess disability across the three domains of work/school, social life, and family life, with each item scored from 0 (not at all) to 10 (very severely), with a summarization of the 3 items to evaluate global functioning. The Global Functional Impairment Score is a total score score that ranges from 0 (unimpaired) to 30 (highly impaired), and was used to derived the mean change from baseline to endpoint.
Time Frame: Baseline, 12 weeks
Population: Intent to Treat. Data based on number of subjects enrolled at Week 0: Duloxetine N=362, SSRI N=370; and Week 12: Duloxetine N=270, SSRI N=283
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 270 | 283
units on a scale | -13.56 (0.53) | -11.53 (0.52)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis

15. Secondary Outcome: Change From Baseline in SDS Work/School Item Score at 12-Week Endpoint (Functional Outcome Measure)
Description: The SDS is completed by the participant and Item 1 is used to assess the effect of the participant's symptoms on their work/school schedule. Scores range from 0 to 10 with higher values indicating greater disruption in the participant's work/school life.
Time Frame: Baseline, 12 Weeks
Population: Intent to Treat. Data based on number of subjects enrolled at Week 0: Duloxetine N=260,SSRI N=267; and Week 12: Duloxetine N=182, SSRI N=192
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 182 | 192
units on a scale | -4.52 (0.22) | -3.85 (0.21)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); Repeated Measures Analysis. Treatment comparisons will include the contrast between treatment groups at endpoint; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis

16. Other Pre Specified Outcome: Change From Baseline in World Health Organization Health and Work Performance Questionnaire, Clinical Trials 7-Day Version (HPQ), Dollars of Income Lost Due to Work Presenteeism (WP)Score, at Week-12 Endpoint
Description: WP score was calculated by taking midpoint of annual before-tax income reported on HPQ. A multiplier of 1.25 produced estimated direct & indirect (i.e. benefits) income. Annual hours expected to work were calculated from expected daily work hours, multiplied by 236 days. Hourly, indirect income was total direct + indirect income, divided by # of expected annual work hours. Indirect hours lost annually for WP=hours expected to be worked annually times WP percent, times hourly rate=dollars earned, and then subtracted from total direct + indirect income=dollars lost annually due to WP.
Time Frame: Baseline, 12 Weeks
Population: Intent to Treat. Last Observation Carried Forward.
Measure: Least Squares Mean (Standard Error); unit: dollars
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 130 | 132
dollars | 7250.93 (954.77) | 5074.09 (957.77)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); Test type: Superiority or Other; p = 0.07, ANCOVA — Between group P-value

17. Other Pre Specified Outcome: Change From Baseline in World Health Organization Health and Work Performance Questionnaire, Clinical Trials 7-Day Version (HPQ), Dollars of Income Lost Due to Work Absenteeism Score at Week-12 Endpoint
Description: Self-administered assessment used to determine a participant's work performance in terms of employment status, absenteeism if employed, productivity while at work, usual occupation, and annual income. Tool assesses the potential impact of change in depressive symptoms on work productivity and its associated employer costs. Scale ranges from 0 to 100% of work days in past 30 days. Absenteeism and presenteeism were combined into a measure of total lost work performance by adding absenteeism to the value ([100-absenteeism] × [100-presenteeism]). Mean change baseline to endpoint.
Time Frame: Baseline, 12 weeks
Population: Intent to Treat. Last Observation Carried Forward.
Measure: Least Squares Mean (Standard Error); unit: dollars
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 134 | 142
dollars | -3978.98 (1708.92) | -1932.46 (1689.85)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); Test type: Superiority or Other; p = 0.34, ANCOVA — Between group P-value

18. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Family/Home Item Score at Week-12 Endpoint (Functional Outcome Measure)
Description: The SDS is completed by the participant and Item 3 is used to assess the effect of the participant's symptoms on their family life/home responsibilities. Scores range from 0 to 10 with higher values indicating greater disruption in the participant's family life/home responsibilities.
Time Frame: Baseline, 12 Weeks
Population: Intent to Treat. Data based on number of subjects enrolled at Week 0: Duloxetine N=363, SSRI N=370; and Week 12: Duloxetine N=271, SSRI N=283
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 271 | 283
units on a scale | -4.51 (0.19) | -3.94 (0.18)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); Repeated Measures Analysis. Treatment comparisons will include the contrast between treatment groups at endpoint; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis

19. Secondary Outcome: Change From Baseline in SDS Social Item Score at 12-Week Endpoint (Functional Outcome Measure)
Description: The SDS is completed by the participant and is used to assess the effect of the participant's symptoms on their work/social/family life. Total scores range from 0 to 30 with higher values indicating greater disruption in the participant's work/social/family life.
Time Frame: Baseline, 12 Weeks
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 270 | 283
units on a scale | -4.69 (0.18) | -4.04 (0.18)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); Repeated Measures Analysis. Treatment comparisons will include the contrast between treatment groups at endpoint; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis

20. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Week-12 Endpoint
Description: Mean change from baseline to endpoint in systolic blood pressure
Time Frame: Baseline, 12 Weeks
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: millimeters of mmercury (mmHg)
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 274 | 285
millimeters of mmercury (mmHg) | 0.58 (0.69) | 0.55 (0.68)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); Repeated Measures Analysis. Treatment comparisons will include the contrast between treatment groups at endpoint; Test type: Superiority or Other; p = 0.97, Mixed Models Analysis

21. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Week-12 Endpoint
Description: Mean change from baseline to endpoint in diastolic blood pressure
Time Frame: Baseline, 12 Weeks
Population: Intent to Treat. Data based on number of subjects enrolled at Week 0: Duloxetine N=367, SSRI N=371: and Week 12: Duloxetine N=274, SSRI N=285
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 274 | 285
mmHg | -0.14 (0.48) | 0.45 (0.46)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); Repeated Measures Analysis. Treatment comparisons will include the contrast between treatment groups at endpoint; Test type: Superiority or Other; p = 0.32, Mixed Models Analysis

22. Other Pre Specified Outcome: Change From Baseline in World Health Organization Health and Work Performance Questionnaire, Clinical Trials 7-Day Version (HPQ), Absenteeism at 12-Week Endpoint
Description: Self-administered assessment used to determine a subject's work performance in terms of employment status, absenteeism if employed, productivity while at work, usual occupation, and annual income. Tool assesses the potential impact of change in depressive symptoms on work productivity and its associated employer costs. Defined on a 0-100 scale for the percentage of work days the respondent missed in the past 30 days. Absolute absenteeism: actual hours worked minus expected hours equals number of missed work days. Mean change baseline to endpoint is reported.
Time Frame: Baseline, 12 Weeks
Population: Intent to Treat. Last Observation Carried Forward.
Measure: Least Squares Mean (Standard Error); unit: hours lost per week
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 137 | 146
hours lost per week | -9.56 (5.14) | 0.41 (5.05)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); Transformed absolute score; Test type: Superiority or Other; p = 0.12, ANCOVA — Between group P-value

23. Other Pre Specified Outcome: Change From Baseline in World Health Organization Health and Work Performance Questionnaire, Clinical Trials 7-Day Version (HPQ), Presenteeism Score, at Week-12 Endpoint
Description: Self-administered assessment used to determine a participant's work performance (employment status, absenteeism if employed, productivity while at work, usual occupation, & annual income). Tool assesses the potential impact of change in depressive symptoms on work productivity & its associated employer costs using a 0-100 scale in which 0 meant doing no work at all on days spent at work and 100 meant performing at the level of a top worker. Absolute presenteeism: difference between "score for self" and "score for average worker in same job". Mean change baseline to endpoint is reported.
Time Frame: Baseline, 12 Weeks
Population: Intent to Treat. Last Observation Carried Forward.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 136 | 139
units on a scale | 24.56 (2.14) | 20.73 (2.11)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); Transformed Absolute Score; Test type: Superiority or Other; p = 0.16, ANCOVA — Between group P-value

24. Secondary Outcome: Change From Baseline in Pulse Rate at Week-12 Endpoint
Description: Mean change from baseline to endpoint in pulse rate
Time Frame: Baseline, 12 Weeks
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 274 | 285
beats per minute (bpm) | 2.74 (0.58) | 0.47 (0.57)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); Repeated Measures Analysis. Treatment comparisons will include the contrast between treatment groups at endpoint; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis

25. Secondary Outcome: Change From Baseline in Weight at Week-12 Endpoint
Description: Mean change from baseline to endpoint in weight
Time Frame: Baseline, 12 Weeks
Population: Intent to Treat. Data based on number of subjects enrolled at Week 0: Duloxetine N=366, SSRI N=370; and Week 12: Duloxetine N=273, SSRI N=284
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | Duloxetine | Selective Serotonin Reuptake Inhibitor (SSRI)
Number analyzed (Participants) | 273 | 284
kilograms (kg) | -0.32 (0.18) | -0.17 (0.18)
Statistical Analysis 1: Comparison: Duloxetine vs Selective Serotonin Reuptake Inhibitor (SSRI); Repeated Measures Analysis. Treatment comparisons will include the contrast between treatment groups at endpoint; Test type: Superiority or Other; p = 0.53, Mixed Models Analysis

ADVERSE EVENTS:
Groups:
- Duloxetine: 30-120 mg orally daily for 12 weeks
- Citalopram: 20-40 mg orally daily for 12 weeks
- Fluoxetine: 20-80 mg orally daily for 12 weeks
- Paroxetine: 20-50 mg orally daily for 12 weeks
- Sertraline: 50-200 mg orally daily for 12 weeks
Arm/Group | Duloxetine | Citalopram | Fluoxetine | Paroxetine | Sertraline
Serious Adverse Events (participants affected / at risk) | 4/372 | 2/157 | 1/57 | 1/45 | 2/119
Other Adverse Events (participants affected / at risk) | 277/372 | 112/157 | 47/57 | 36/45 | 86/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=372) | Citalopram (N=157) | Fluoxetine (N=57) | Paroxetine (N=45) | Sertraline (N=119)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Temporal lobe epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=372) | Citalopram (N=157) | Fluoxetine (N=57) | Paroxetine (N=45) | Sertraline (N=119)
Constipation (Gastrointestinal disorders) | 33 (35) | 8 (8) | 1 (2) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 36 (41) | 17 (18) | 10 (10) | 3 (3) | 18 (20)
Dry mouth (Gastrointestinal disorders) | 66 (67) | 16 (16) | 11 (11) | 4 (4) | 13 (13)
Nausea (Gastrointestinal disorders) | 63 (70) | 17 (18) | 8 (9) | 8 (8) | 15 (16)
Fatigue (General disorders) | 27 (28) | 10 (10) | 2 (3) | 8 (8) | 3 (3)
Nasopharyngitis (Infections and infestations) | 11 (11) | 5 (5) | 1 (2) | 4 (4) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 8 (8) | 2 (2) | 1 (1) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 18 (18) | 5 (5) | 4 (4) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (5) | 3 (3) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (13) | 4 (4) | 3 (3) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 23 (26) | 4 (4) | 1 (1) | 5 (5) | 7 (7)
Headache (Nervous system disorders) | 55 (62) | 16 (18) | 8 (11) | 6 (6) | 16 (19)
Somnolence (Nervous system disorders) | 27 (27) | 11 (11) | 2 (2) | 3 (3) | 3 (3)
Anorgasmia (Psychiatric disorders) | 4 (4) | 3 (3) | 1 (1) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 25 (25) | 3 (3) | 8 (9) | 3 (3) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 12 (13) | 1 (1) | 3 (3) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days